CLINICAL TRIAL: NCT01904929
Title: Evaluation of the Psychometric Properties of the 400m-walk-test at a Self-selected Speed (400m WT) for Stable Coronary Patients
Brief Title: The 400m-walk-test for Stable Coronary Patients
Acronym: TML 400 m
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CASILLAS TML 400m 2013
Record Dates: First submitted 2013-07-08; First posted 2013-07-22 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Chronic Coronary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reconditioning in the effort (Experimental)
  Interventions: Other: Walk-tests

INTERVENTIONS:
Other: Walk-tests — Patients will make a 6-minute-walk-test, the 400m-walk-test and a 200m-fast walk test. These first 2 tests (TM6min and TML400m) will be made in an order determined by randomization.
  This series of test will be repeated 72 hours later for the study reproducibility.
  It will be followed by a phase of rest of 15 min and a test of effort on travelator, according to the protocol of " modified Bruce " in moderation of portable VO2.

SUMMARY:
The objective of this project is to clarify and improve the efficiency of the standardized walk-test in Cardiovascular Rehabilitation. The psycho-metric properties of the 400m walk test at a self-selected speed will be evaluated. Such tests, made at a self-selected ("comfortable", "free") speed particularly assess the endurance capacities. The results of the physiological measurements during the tests will be compared with those of TM6min of Test of Fast Walking of 200m (TMR200m) and a maximal treadmill exercise. Stable coronary patients, aged over 55 years old, will be included.

This study should permit a simplification and a better understanding of the clinical-use of walk tests. In the future, two kinds of tests might be proposed with different distances, 1- 200m-fast-walking-test aimed to evaluate the performance closed to the maximum capacity, 2- self-selected-walk-test on a doubled distance (400m) aimed to evaluate the aerobic capacities of the adaptation of the body in response to effort.

ELIGIBILITY:
Inclusion Criteria:

* Patient received enlightened information on research.
* Patient affiliated to healthcare insurance.
* Patients who agreed to participate in the study.
* Patient male or female aged 55 or more.
* Chronic coronary patient who completed his rehabilitation program.
* Patient able to understand simple orders.
* Indication of outpatient rehabilitation in coronary angioplasty + stenting, surgical coronary revascularization (coronary artery bypass), acute coronary syndrome (STEMI or NO STEMI) or stable angina suites.

Exclusion Criteria:

* Patient under guardianship or tutelage
* Arrhythmia or pace maker (making criterion heart rate unusable).
* Congestive heart failure with left ventricular ejection fraction <45% measured by trans-thoracic echocardiography according to Simpson's method or assay plasma N-terminal pro-brain natriuretic peptide (NT-pro-BNP-3) times the values used in healthy subjects by the analytical laboratory of the University Hospital of Dijon.
* Severe obstructive cardiomyopathy.
* Aortic valve.
* Thrombus intra cavitary.
* Severe pulmonary hypertension (> 70 mm Hg).
* History of venous thromboembolism in the last 3 months.
* Heart Transplantation.
* Chronic motor impairments associated with neurological (e.g. sequelae of stroke, impaired balance and coordination) or musculoskeletal origin (e.g., osteoarthritis, osteoarthritis), because the secondary functional impairment will limit the ability to work predominantly in relation to the adaptation to stress.
* Severe medical disorder associated to a significantly alteration of the functional capacity (respiratory failure, metabolic disorders such as non-stabilized progressive renal failure) and involving the vital prognosis in the short or medium term (neoplasIC pathology progressive, systemic disease, non-stabilized).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Measurement of intra-class correlation coefficient (ICC) | 3 days
  Measurement between:
  * 1) The Maximal consumption of oxygen (VO2) uptake during the 400m-walk-test (TML400m) and the VO2 value at the first aerobic threshold measured during graded maximal exercise on treadmill.
  * 2) the heart rate during TML400 and the heart rate value at the first aerobic threshold measured during graded maximal exercise on treadmill.
  These ICC will be also assessed, during a 6-minute-walk-test and a 200m-fast walk test compared to the maximal graded test.

SECONDARY OUTCOMES:
A variance analysis (ANOVA) | 3 days
  To determine differences between the different measures performed in the VO2 tests. If a significant difference is found, a post-hoc LSD(Least Significant Difference)test types will be conducted to classify the variables.
Univariate analysis | 3 days
  To search for potential relationships between the maximum heart rate and the following variables: age, height, weight, BMI, HRrest (resting heart rate), FC6mn (heart rate at 6 minutes), T6mn (T=6 minutes), FCT200, TMR200 (Test of fast walking of 200m), and TML400. To select the variables of interest, we will use a stepwise method using algorithms available in the NCSS 2004 software (Statistical software).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon, Dijon, France